CLINICAL TRIAL: NCT05831176
Title: A Phase 2, 2-Part, Open-Label, Single-Arm Study to Investigate the Efficacy and Safety of Dupilumab in Adult and Adolescent Patients With Eosinophilic Gastritis With or Without Eosinophilic Duodenitis
Brief Title: A Study to Learn How Well Dupilumab Works in Adult and Adolescent Participants With Eosinophilic Gastritis With or Without Eosinophilic Duodenitis and the Side Effects it May Have
Acronym: ENGAGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-EGE-2213; 2022-500795-62-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Gastritis (EoG); Eosinophilic Duodenitis (EoD); Eosinophilic Gastrointestinal Disease (EGID); Eosinophilic Gastroenteritis
Keywords: Eosinophilic Gastritis (EoG) with or without Eosinophilic Duodenitis (EoD)
MeSH Terms: conditions — Eosinophilic enteropathy; Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab (Experimental): Part A: Treatment Period Part C: Extended Treatment Period
  Eligible participants from Part A will enter Part C
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Administered as described in the protocol
  Other Names: DUPIXENT®; REGN668; SAR231893

SUMMARY:
This study is researching an experimental drug called dupilumab. The study is focused on participants with active eosinophilic gastritis (EoG) with or without eosinophilic duodenitis (EoD). Participants with EoD only are not eligible for enrollment. EoG and EoD are uncommon, persistent, allergic/immune diseases in which eosinophils (a type of white blood cell) gather in large numbers in the stomach and small intestine and cause inflammation and damage.

The aim of the study is to evaluate the effect of dupilumab on relieving EoG (with or without EoD) symptoms and reducing inflammation in the stomach and, if applicable, small intestine in adults and adolescents aged 12 years and older after at least 24 weeks (about 6 months) and up to 52 weeks (1 year) of treatment.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

DETAILED DESCRIPTION:
This study has 2 parts and a 12-week (about 3 months) Follow-up Period for all participants

* Part A is an open-label treatment period lasting up to 24 weeks (up to 6 months). "Open-label" means that you and the study doctors and the staff staff will know that you are taking the study drug
* Part C is an open-label extended treatment period lasting up to 28 weeks (about 7 months). "Extended Treatment Period" means that you will take the study drug for an additional 28 weeks after finishing Part A if you are eligible to take part in this part of the study

ELIGIBILITY:
Key Inclusion Criteria:

1. Adolescent participants will only be enrolled at study sites in countries/regions as permitted by local regulatory authorities and ethic committees (ECs)
2. Documented endoscopic biopsy supporting a pathologic diagnosis of Eosinophilic gastritis (EoG) at least 3 months prior to screening
3. Screening endoscopic biopsies with a demonstration of eosinophilic infiltration for a diagnosis of EoG, as defined in the protocol
4. Completed at least 11 of 14 days of EoG/EoD-SQ eDiary data entry in the 2 weeks prior to the baseline visit
5. History (by participant report) of at least 2 episodes of EoG (with or without EoD) symptoms per week in 8 weeks before screening, as defined in the protocol
6. An average TSS of ≥ 20 calculated using data collected via the EoG/EoD-SQ eDiary per week for the 2 weeks prior to baseline. An average severity score of ≥4 (on a scale of 0-10) per week for the 2 weeks prior to baseline for at least 2 of the 6 symptoms, as defined in the protocol.

Key Exclusion Criteria:

1. Body weight less than 40 kg at screening
2. Prior participation in a dupilumab clinical trial, or past or current treatment with dupilumab
3. Helicobacter pylori infection
4. Any esophageal stricture unable to be passed with a standard, diagnostic, upper endoscope or any critical esophageal stricture that requires dilation at screening
5. History of achalasia, Crohn's disease, eosinophilic colitis, ulcerative colitis, celiac disease, and prior gastric or duodenal surgery, as defined in the protocol
6. Other causes of gastric and, if applicable, duodenal eosinophilia or the following conditions: eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome) or hyper-eosinophilic syndrome
7. History of bleeding disorders, esophageal or gastric varices that, in the opinion of the investigator, would put the participant at undue risk for significant complications from an endoscopy procedure
8. Initiation or change of a food-elimination diet regimen or re-introduction of a previously eliminated food group in the 4 weeks prior to the screening visit. Participants on a food-elimination diet must remain on the same diet throughout the study
9. Planned or anticipated use of any prohibited medications and procedures during the study
10. Planned or anticipated major surgical procedure during the study
11. Receiving tube feeding or parenteral nutritional at screening

NOTE: Other Protocol Defined Inclusion / Exclusion Criteria Apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Percent change in peak gastric eosinophil count eosinophils/high power field (eos/hpf) | Baseline up to 24 Weeks

SECONDARY OUTCOMES:
Percent change in peak gastric eosinophil count eosinophils/high power field (eos/hpf) | Baseline up to 52 Weeks
Proportion of participants achieving a peak gastric eosinophil count of ≤20 eos/hpf | Up to 52 Weeks
Proportion of participants achieving a peak gastric eosinophil count of ≤30 eos/hpf | Up to 52 Weeks
Proportion of participants achieving both a peak gastric eosinophil count of ≤20 eos/hpf and a peak duodenal eosinophil count of ≤30 eos/hpf | Up to 52 Weeks
Proportion of participants achieving a peak duodenal eosinophil count of ≤30 eos/hpf | Up to 52 Weeks
  Assessed for only those with duodenal involvement
Absolute change in the EoG/EoD-SQ Total Symptom Score (TSS) | Baseline up to 52 Weeks
  EoG/EoD-SQ is a PRO collected daily via an eDiary. Symptoms are assessed using an 11-point numerical rating scale (0 through 10). Higher scores indicate a higher symptom burden. Symptom scores are summed on each day with a maximum daily score of 60. The TSS is calculated by averaging daily sum scores over 7 days, with a maximum TSS of 60.
Percent change in the EoG/EoD-SQ TSS | Baseline up to 52 Weeks
Percent change in peak duodenal tissue eosinophil count (eos/hpf) | Baseline up to 52 Weeks
  Assessed for only those with duodenal involvement
Absolute change in EoG scores from the EoG Histology Scoring System (EoGHSS) | Baseline up to 52 Weeks
  EoGHSS scores evaluate 11 features of gastric tissue. Total score is the sum of features scores divided by the maximum possible score for the biopsy. Total scores range from 0 - 1.
Change in frequency of diarrhea episodes | Baseline up to 52 Weeks
  Assessed for only those with diarrhea at baseline
Change in frequency of vomiting episodes | Baseline up to 52 Weeks
  Assessed for only those with vomiting at baseline
Change in the Normalized Enrichment Scores (NES) for the type 2 inflammation transcriptome signature | Baseline up to 52 Weeks
  Assessed on gastric tissue
  Normalized Enrichment Score (NES) reflects the degree to which the activity level of a set of transcripts is overrepresented at the extremes (top or bottom) of the entire ranked list of transcripts within a sample and is normalized by accounting for the number of transcripts in the set.
Change in the NES for the type 2 inflammation transcriptome signature | Baseline up to 52 Weeks
  Assessed on duodenal tissue from participants with EoD
  NES reflects the degree to which the activity level of a set of transcripts is overrepresented at the extremes (top or bottom) of the entire ranked list of transcripts within a sample and is normalized by accounting for the number of transcripts in the set.
Change in the NES for the EoG disease (EoG diagnostic panel (EGDP]) transcriptome signature | Baseline up to 52 Weeks
  Assessed on gastric tissue
  NES reflects the degree to which the activity level of a set of transcripts is overrepresented at the extremes (top or bottom) of the entire ranked list of transcripts within a sample and is normalized by accounting for the number of transcripts in the set.
Proportion of participants who receive rescue medications or procedures | Up to 52 Weeks
Incidence of treatment-emergent adverse events (TEAEs) | Up to 52 Weeks
  A TEAE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Incidence of treatment-emergent serious adverse events (SAEs) | Up to 52 Weeks
  An SAE is any untoward medical occurrence that at any dose:
  * Results in death - includes all deaths, even those that appear to be completely unrelated to study drug (eg, a car accident in which a patient is a passenger)
  * Is life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event
Incidence of treatment-emergent adverse events of special interest (AESIs) | Up to 52 Weeks
  An AESI (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it
Incidence of TEAEs leading to permanent discontinuation of study treatment | Up to 52 Weeks
  A TEAE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Incidence of anti-drug antibody (ADA) | Up to 52 Weeks
  Immunogenicity will be characterized per drug molecule by ADA status
Titer of ADA | Up to 52 Weeks
  Immunogenicity will be characterized per drug molecule by ADA status
Incidence of neutralizing antibody (NAb) to dupilumab | Up to 52 Weeks
  Immunogenicity will be characterized per drug molecule by NAb status
Concentrations of functional dupilumab in serum at each assessment time point | Baseline up to 64 Weeks
  The concentrations of functional dupilumab over time will be summarized by descriptive statistics by study arm for the overall population and for adolescent patients.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (53):
- United States (36):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Om Research LLC, Apple Valley, California
  - Scripps Clinic, La Jolla, California
  - Om Research LLC, Lancaster, California
  - University of California - Los Angeles (UCLA), Los Angeles, California
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - GastroIntestinal BioSciences, Los Angeles, California
  - United Medical Doctors, Murrieta, California
  - Ucsf Medical Center (Benioff Childrens Hospital), San Francisco, California
  - University of Colorado Anschutz Health Science Building (AHSB) CU Research Pharmacy, Aurora, Colorado
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - UConn Health, Farmington, Connecticut
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University Of Kansas, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center (BIDMC) Harvard Medical School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - MNGI Digestive Health P.A., Plymouth, Minnesota
  - Mayo Clinic Hospital Rochester, Rochester, Minnesota
  - Advanced Research Institute, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Northwell Health, Great Neck, New York
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH), New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - ESI Medical Research, PLLC, Kinston, North Carolina
  - University of Cincinnati Medical Center-Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - The Oregon Clinic - Gastroenterology East, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - TDDC dba GI Alliance Research, Mansfield, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Home Health Company, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- Stollery Children's Hospital - University of Alberta, Edmonton, Alberta, Canada
- Italy (7):
  - Humanitas Research Hospital, Rozzano, Milan
  - AOOR Villa Sofia/Cervello, Palermo, Sicily
  - U.O. Di Ematologia-Azienda Policlinico Consorziale, Ospedaliero-Universitaria, Ospedale, Bari
  - Fondazione Serena Onlus - Azienda Ospedaliera Niguarda Ca' Granda - Centro Clinico Nemo (Neuro Muscular Omnicentre), Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale S Giovanni Calibita Fatebenefratelli Isola Tiberina, Roma
  - University of Rome - Pediatric Gastroenterology and Liver Unit, Rome
- Japan (9):
  - Iizuka Hospital, Iizuka, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Kure Kyosai Hospital, Kure, Hiroshima
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji, Hyōgo
  - Kobe University Graduate School of Medicine, Kobe, Hyōgo
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken
  - Toranomon Hospital, Minato-ku, Tokyo
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Sia T, Bacchus L, Tanaka R, Khuda R, Mallik S, Leung J. Dupilumab Can Induce Remission of Eosinophilic Gastritis and Duodenitis: A Retrospective Case Series. Clin Transl Gastroenterol. 2024 Jan 1;15(1):e00646. doi: 10.14309/ctg.0000000000000646. PMID 37753954